CLINICAL TRIAL: NCT01188603
Title: Evaluation of Single Dose and Steady State Pharmacokinetics of Flibanserin Postmenopausal Women With Hypoactive Sexual Desire Disorder
Brief Title: Pharmacokinetics of Flibanserin in Postmenopausal Women With Hypoactive Sexual Desire Disorder (HSDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511.146
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2012-04-10 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- flibanserin (Experimental): flibanserin 100 mg dose every evening
  Interventions: Drug: flibanserin 100 mg dose every evening

INTERVENTIONS:
Drug: flibanserin 100 mg dose every evening — all subjects receive flibanserin

SUMMARY:
This trial examines the way flibanserin is metabolized in postmenopausal women with Hypoactive Sexual Desire Disorder.

ELIGIBILITY:
Inclusion criteria:

1. Patients must be in a stable, monogamous heterosexual relationship for at least one year.
2. Patients must have a primary diagnosis of Hypoactive Sexual Desire Disorder for at least six months.
3. Patients must be naturally postmenopausal women of any age with at least one ovary.
4. Patients may participate whether or not they are currently taking systemic hormone therapy provided the therapy was not prescribed for treatment of low sexual desire. Hormone therapy must be at a stable dose for at least six months.

Exclusion criteria:

1. Patients with a history of drug dependence or abuse within the past twelve months.
2. Patients who have been previously treated with flibanserin.
3. Patients who have sexual dysfunctions other than Hypoactive Sexual Desire Disorder, such as: Sexual Aversion Disorder, Substance-Induced Sexual Dysfunction, Dyspareunia, Vaginismus, Gender Identity Disorder,Paraphilia, or Sexual Dysfunction due to a general medical condition.
4. Patients who indicate that their sexual partner has inadequately treated organic or psychosexual dysfunction that could interfere with a patients response to treatment.
5. Patients whose sexual function was impaired, in the investigators opinion, by abdominal or vaginal hysterectomy, oophorectomy or any other pelvic, vaginal, or urologic surgery.
6. Patients with pelvic pain, pelvic inflammatory disease, endometriosis, urinary tract or vaginal infection/vaginitis, cervicitis, interstitial cystitis, vulvodynia, symptomatic vaginal atrophy or any other gynecological pathology requiring further evaluation.
7. Patients with a history of unexplained vaginal bleeding within the past twelve months.
8. Patients with a history of Major Depressive Disorder within six months prior to Screening; ; active suicidal ideation with intent in the past ten years or suicidal behavior at any time.
9. Patients with a history of any other psychiatric disorder that could impact sexual function, increase risks to patient safety, or impair patient compliance. Such disorders include but are not limited to bipolar disorder, psychotic disorders, severe anxiety, eating disorders, and antisocial personality disorders.
10. Clinically significant electrocardiogram abnormalities at Screening.
11. Patients with a history of dementia or other neurodegenerative disease; organic brain disease; stroke; transient ischemic attacks; multiple sclerosis; spinal cord injury; brain surgery; significant brain trauma; peripheral neuropathy; and epilepsy.
12. Patients with ongoing hepatic impairment (cirrhosis, hepatic tumor, or other hepatic disease); peptic ulcer within six months prior to Screening; elevated liver enzymes ; inflammatory bowel disease; gastrointestinal bleeding within two months prior to Screening; Patients who have had bariatric surgery for obesity.
13. Patients with a history of angina; atherosclerotic cardiovascular disease; congestive heart failure; cardiomyopathy; symptomatic cardiac valve disease; arrhythmia; hypertension.
14. Patients with a history of renal failure; known history of chronic glomerulonephritis.
15. Patients with a history of chronic obstructive pulmonary disease, chronic bronchitis, or asthma not well controlled with medication taken twice daily or less.
16. Patients with a history of gonadotrophic hormone disorders or uncontrolled diabetes mellitus.
17. Uncorrected hypothyroidism or hyperthyroidism.
18. Patients with a history of uncontrolled glaucoma.
19. Patients with known Human Immunodeficiency Virus infection, Acquired Immunodeficiency Syndrome, other clinically significant immunological disorders or auto-immune disorders such as lupus or scleroderma.
20. Patients with a history of any cancer within the past ten years, other than non-invasive, previously resected basal cell carcinoma of the skin.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sprout Pharmaceuticals, Study Chair — Sprout Pharmaceuticals
Locations (4):
- United States (4):
  - 511.146.01003 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.146.01005 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 511.146.01001 Boehringer Ingelheim Investigational Site, Kalamazoo, Michigan
  - 511.146.01004 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Flibanserin: 100mg Flibanserin administered orally once daily
Period: Overall Study
Arm/Group | Flibanserin
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Flibanserin
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 28.25 (5.31)

OUTCOME MEASURES:

1. Primary Outcome: Flibanserin: Area Under the Curve; AUC_0-∞
Description: Geometric mean of the AUC_0-∞ of Flibanserin
Time Frame: 8 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Flibanserin
Number analyzed (Participants) | 22
ng*h/mL | 2570 (73.0)

2. Primary Outcome: Flibanserin: AUC τ,ss
Description: Geometric mean of the AUC τ,ss of Flibanserin
Time Frame: 8 days
Population: All patients with values for the area under the concentration-time curve of the analyte in plasma over a dosing interval τ at steady state (AUC τ,ss)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Flibanserin
Number analyzed (Participants) | 24
ng*h/mL | 3000 (60.9)

3. Primary Outcome: Flibanserin: Cmax (Peak Concentration)
Description: Geometric mean of the Cmax of Flibanserin
Time Frame: 8 days
Population: All patients with values for the maximum concentration of Flibanserin in plasma after single dose (Cmax)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Flibanserin
Number analyzed (Participants) | 22
ng/mL | 298 (56.4)

4. Primary Outcome: Flibanserin: Cmax,ss
Description: Geometric mean of the Cmax,ss of Flibanserin
Time Frame: 8 days
Population: All patients with values for the maximum concentration of Flibanserin in plasma after single dose at steady state (Cmax,ss)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Flibanserin
Number analyzed (Participants) | 24
ng/mL | 406 (60.7)

5. Primary Outcome: Flibanserin: Tmax,ss
Description: Median of the tmax,ss of Flibanserin
Time Frame: 8 days
Population: All patients with values for the time from dosing to the maximum measured concentration of flibanserin in plasma after single dose at steady state (tmax,ss)
Measure: Median (Full Range); unit: h
Arm/Group | Flibanserin
Number analyzed (Participants) | 24
h | 1.50 (0.500;3.00) [0.500 to 3.00]

ADVERSE EVENTS:
Arm/Group | Flibanserin
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 13/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flibanserin (N=24)
Constipation (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Sprout Pharmaceuticals publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.